CLINICAL TRIAL: NCT02385110
Title: Alemtuzumab or Tocilizumab in Combination With Etoposide and Dexamethasone for the Treatment of Adult Patients With Hemophagocytic Lymphohistiocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0989; NCI-2015-00526 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Leukemia
Keywords: Leukemia; Hemophagocytic lymphohistiocytosis; HLH; Alemtuzumab; CAMPATH-1H; Campath; Etoposide; VePesid; Dexamethasone; Decadron; Methotrexate; Phone call
MeSH Terms: conditions — Leukemia; Lymphohistiocytosis, Hemophagocytic | interventions — Alemtuzumab; Etoposide; Dexamethasone; Calcium Dobesilate; Methotrexate; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Alemtuzumab + Etoposide + Dexamethasone (Experimental): Induction Phase: Participants receive Alemtuzumab daily on Days 1 - 4 with weekly Etoposide, and Dexamethasone by vein on Days 1-7 during the 8-weeks. Participants with central nervous system involvement receive intrathecal methotrexate 12 mg once a week for 5 weeks.
  Dexamethasone by vein on Days 1-7 of the induction phase.
  Maintenance Phase: Starts Post Induction Phase for16 weeks. Participants receive Alemtuzumab once every 4 weeks and Dexamethasone three times per week. Participants who have evidence of budding relapse may revert back to receiving Etoposide.
  If participant responds to study drugs, they will receive a phone call by study staff every 3 - 6 months for up to 5 years after completion of treatment. Each call will last about 5-10 minutes.
  Interventions: Drug: Alemtuzumab; Drug: Etoposide; Drug: Dexamethasone; Drug: Methotrexate; Behavioral: Phone Call
- Group 2: Etoposide + Dexamethasone + Tocilizumab (Experimental): Induction Phase: Participants receive Tocilizumab by vein over 60 minutes on Day 1 or Day 2. Participants receive Alemtuzumab daily on Days 1 - 4 with weekly Etoposide and Dexamethasone by vein on Days 1-7 during the 8-weeks. Participants with central nervous system involvement receive intrathecal methotrexate 12 mg once a week for 5 weeks.
  Maintenance Phase: Starts Post Induction Phase and will last 16 weeks. Tocilizumab not given in the Maintenance Phase. Dexamethasone three times per week.
  If participant responds to study drugs, they will receive a phone call by study staff every 3 - 6 months for up to 5 years after completion of treatment. Each call will last about 5-10 minutes
  Interventions: Drug: Alemtuzumab; Drug: Etoposide; Drug: Dexamethasone; Drug: Methotrexate; Behavioral: Phone Call; Drug: Tocilizumab

INTERVENTIONS:
Drug: Alemtuzumab — Group 1 and 2 Induction Phase: Alemtuzumab total dose of 1.0 mg/kg subcutaneously or by vein over 4 days (days 1-4) during the 8 week induction phase. Day 1 0.1 mg/kg, Day 2 0.3 mg/kg, Day 3 0.3 mg/kg, Day 4 0.3 mg/kg.
  Group 1 Maintenance Phase: 0.2 mg/kg once every 4 weeks for 6 weeks.
  Other Names: CAMPATH-1H; Campath
Drug: Etoposide — Induction Phase: 150 mg/m2 given by vein once a week for 8 weeks.
  Maintenance Phase: Participants who have evidence of refractory disease or budding relapse during the maintenance phase may revert back to receiving Etoposide.
  Other Names: VePesid
Drug: Dexamethasone — Induction Phase: 10 mg/m2 for 1 week followed by Dexamethasone 5 mg/m2 for 2 weeks followed by Dexamethasone 2.5 mg/m2 for 2 weeks followed by Dexamethasone 1.25 mg/m2 for 2 weeks.
  Maintenance Phase: 1.25 mg/m2 by mouth three times a week for 16 weeks.
  Other Names: Decadron
Drug: Methotrexate — Participants with central nervous system involvement receive intrathecal methotrexate 12 mg once a week for 5 weeks during the Induction Phase.
Behavioral: Phone Call — If participant responds to study drugs, they will receive a phone call by study staff every 3 - 6 months for up to 5 years after completion of treatment. Each call will last about 5-10 minutes.
Drug: Tocilizumab — Induction Phase: Tocilizumab at 4 to 8 mg/kg by vein. Day 1 0.1 mg/kg,Day 2 0.3 mg/kg, Day 3 0.3 mg/kg, Day 4 0.3 mg/kg.
  Arms: Group 2: Etoposide + Dexamethasone + Tocilizumab

SUMMARY:
The goal of this clinical research study is to compare the effect of adding either alemtuzumab or tocilizumab to the drug combination of etoposide and dexamethasone in controlling HLH. The safety of the drug combinations will also be studied.

This is an investigational study. Alemtuzumab, etoposide, tocilizumab, and dexamethasone are not FDA approved for the treatment of HLH. Etoposide is FDA approved and commercially available for the treatment of testicular cancer and lung cancer. Alemtuzumab is FDA approved and commercially available for the treatment of chronic lymphocytic leukemia. Dexamethasone is a steroid used to reduce inflammation. Tocilizumab is FDA approved and commercially available for the treatment of arthritis. The combination of alemtuzumab, etoposide, tocilizumab, and dexamethasone to treat HLH is investigational. The study doctor can explain how the drugs are designed to work.

Up to 40 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Treatment:

If you are found to be eligible to take part in this study, your doctor will assign you to either Group 1 or Group 2.

You will receive the study treatment in 2 parts. The first part of the study will last about 8 weeks (Weeks 1-8) and will be called the "induction phase". The second part of the study will start after the induction phase and will last about 16 weeks (Weeks 9-16). This part will be called the "maintenance phase". However, the parts of the study may be longer or shorter depending on if/how the disease responds to the treatment, how the biomarkers react to treatment, and what the doctor thinks is in your best interest.

* If you are in Group 1, you will receive alemtuzumab by vein over 2 hours or through an injection under the skin every day on Days 1-4 of the induction phase and about 1 time every 4 weeks during the maintenance phase.
* If you are in Group 2, you will receive tocilizumab by vein over 60 minutes on Day 1 or Day 2 of the Induction phase. Tocilizumab will not be given in the Maintenance Phase.

Participants in both Groups 1 and 2 will receive etoposide by vein about 1 time each week during the induction phase. You will not receive it in the maintenance phase unless the disease stops responding to the study drugs. At that point, you may begin to receive etoposide again. The study doctor will tell you more about this.

The length of time it takes to infuse the study drugs will be different from patient to patient and will depend on rate of injection. Your doctor will discuss this with you.

Participants in both Groups 1 and 2 will receive dexamethasone by vein on Days 1-7 of the induction phase. After this, you will take pills of dexamethasone every day during the induction phase. In the maintenance phase, you will take these pills 3 times each week with at least a day between each dose (for example, Monday, Wednesday, and Friday).

Your dose of the study drugs may be raised, lowered, and/or delayed if the doctor thinks it is in your best interest.

If the disease involves the central nervous system during the Induction phase, you may receive methotrexate. Methotrexate is given 1 time a week for 5 weeks.

Study Visits:

You will have physical exams on the following days:

* Day 1,
* Every week for the first 4 weeks,
* Every 2 weeks during the next 4 weeks,
* Every 4 weeks during the next 16 weeks, and
* Every 8 weeks after that.

Blood (about 3 tablespoons) will be drawn for routine tests on the following days. During the first 4 weeks, these tests must be performed at MD Anderson. After that, these can be performed at a local clinic:

* Day 1,
* Two (2) times each week for the first 4 weeks,
* Every week for the next 4 weeks,
* Every 2 weeks for the next 16 weeks, and
* Every 4 weeks after that.

You will have a bone marrow aspiration/biopsy 4 weeks after starting the study treatment and then every 4-12 weeks after that.

At any time that the doctor thinks it is needed, you may have additional blood draws or bone marrow aspirations/biopsies to check the status of the disease. If you receive treatment for longer than 24 weeks, the timing of these procedures may be changed if the study doctor thinks it is in your best interest.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Study Visit:

If you are taken off or if you leave the study before you have received treatment for 24 weeks, the following tests and procedures will be performed within 30 days (+/- 7 days) of the last dose of the study drug:

* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a bone marrow aspirate to check the status of the disease.

If you cannot make it to MD Anderson for this visit, these procedures may be done with a local doctor and the records can be forwarded to the study doctor.

Follow-Up:

If you respond to the study drugs, you will be followed every 3-6 months for up to 5 years after completion of treatment. You will be called and asked about how you are doing. Each call will last about 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an IRB-approved informed consent document.
2. Patients must be >/= 18 years of age.
3. • A documentation of diagnosis of hemophagocytic lymphocytosis, either newly diagnosed or relapsed/refractory by the treating physician and the PI in the patients chart. It must be noted that no diagnostic criteria have been established for diagnosis of HLH in adult patients as this was a hitherto poorly identified and considered to be a very rare disease in adults. We have seen an increasing number of cases of HLH at our institution over the last 2 years partly due to referrals and partly due to better understanding of the disease through discussions with our collaborators Dr Kenneth McClain and Dr Carl Allen at TCH (experts in pediatric HLH). Adult HLH seems to occur more frequently post malignancy and has a more fulminant course than pediatric HLH.
4. Continued from No. 3: The diagnostic criteria that have been traditionally used for children (HLH 1991 and HLH 2004) may not adequately diagnose HLH in adults. This is the first adult HLH protocol in the country. In the absence of standard diagnostic guidelines if the patient's symptoms are highly suspicious for HLH and after an adequate work-up to rule out alternate potential alternate etiologies is performed we will treat the patient for HLH as missing the diagnosis is associated with high mortality. These patients will be discussed with the PI (Dr Daver) prior to enrollment in all such cases.
5. Organ function as defined below (unless due to the HLH process): Serum creatinine </= 3.0 mg/dL, Total bilirubin </= 5.0 mg/dL. If organ dysfunction is thought to be related to the HLH process this must be clearly documented in the chart and the patients may be enrolled on study irrespective of creatinine and bilirubin levels.
6. Women of childbearing potential must practice contraception. Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation. Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, prior to study entry and for at least 3 months after the last dose of study drug.
7. Negative urine pregnancy test and/or serum pregnancy test within 7 days of initiation of therapy.
8. Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, prior to study entry and for at least 3 months after the last dose of study drug.

Exclusion Criteria:

1. Pregnant and breast feeding women
2. Any serious/and or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
3. Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: Alemtuzumab + Etoposide + Dexamethasone | Group 2: Etoposide + Dexamethasone + Tocilizumab
Started | 2 | 16
Completed | 1 | 16
Not Completed | 1 | 0
Not completed — Early Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Etoposide + Dexamethasone + Tocilizumab: IInduction Phase: Participants receive Tocilizumab by vein over 60 minutes on Day 1 or Day 2. Participants receive Alemtuzumab daily on Days 1 - 4 with weekly Etoposide and Dexamethasone by vein on Days 1-7 during the 8-weeks. Participants with central nervous system involvement receive intrathecal methotrexate 12 mg once a week for 5 weeks.
  Maintenance Phase: Starts Post Induction Phase and will last 16 weeks. Tocilizumab not given in the Maintenance Phase. Dexamethasone three times per week.
  If participant responds to study drugs, they will receive a phone call by study staff every 3 - 6 months for up to 5 years after completion of treatment. Each call will last about 5-10 minutes
- Total: Total of all reporting groups
Arm/Group | Group 1: Alemtuzumab + Etoposide + Dexamethasone | Group 2: Etoposide + Dexamethasone + Tocilizumab | Total
Number analyzed (Participants) | 2 | 16 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 13 | 15
  >=65 years | 0 | 3 | 3
Age, Continuous [Median (Full Range); unit: years] | 27 [25 to 48] | 54 [31 to 82] | 50 [25 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 2 | 10 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 11 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 16 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response to Alemtuzumab or Tocilizumab in Combination With Etoposide and Dexamethasone for the Treatment of Adult Patients With Hemophagocytic Lymphohistiocytosis
Description: Response is defined as complete response (CR) and/or partial response (PR) and/or parameter improvements (PI). Complete response (CR) is normalization to within institutional normal limits of diagnostic clinical and laboratory abnormalities associated with HLH. In the case of ferritin, normalization OR a 3 fold improvement in the pre-study level will be evidence of complete response, provided the post therapy level is also below 10000 ng/ml. Partial response (PR) is sustained normalization of 3 or more of the diagnostic clinical and laboratory abnormalities noted above (or, with ferritin, improvement as described above) and no apparent progression of other aspects of disease pathology. Parameter improvements (PI) is at least a 25% improvement in two or more quantifiable symptoms and/or laboratory markers from those mentioned above within 8 weeks (+/- 7 days) of initiation of therapy.
Time Frame: 8 weeks
Population: Of the two participants in Group 1, only one participant was evaluable for response. Of the sixteen participants in Group 2, only eight were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Alemtuzumab + Etoposide + Dexamethasone | Group 2: Etoposide + Dexamethasone + Tocilizumab
Number analyzed (Participants) | 1 | 8
Participants | 1 | 8

2. Primary Outcome: Disease Free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: 8 weeks
Population: Of the two participants in Group 1, only one participant was evaluable for response. Of the 16 participants in Group 2, only eight were evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Group 1: Alemtuzumab + Etoposide + Dexamethasone | Group 2: Etoposide + Dexamethasone + Tocilizumab
Number analyzed (Participants) | 1 | 8
Months | 1.9 | 1.9 [0.8 to 5.0]

ADVERSE EVENTS:
Time Frame: Up to 7 years, 3 months
Arm/Group | Group 1: Alemtuzumab + Etoposide + Dexamethasone | Group 2: Etoposide + Dexamethasone + Tocilizumab
All-Cause Mortality (participants affected / at risk) | 1/2 | 7/16
Serious Adverse Events (participants affected / at risk) | 1/2 | 9/16
Other Adverse Events (participants affected / at risk) | 2/2 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Alemtuzumab + Etoposide + Dexamethasone (N=2) | Group 2: Etoposide + Dexamethasone + Tocilizumab (N=16)
Fever (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Alemtuzumab + Etoposide + Dexamethasone (N=2) | Group 2: Etoposide + Dexamethasone + Tocilizumab (N=16)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Catheter Related Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 6 (6)
Fatigue (General disorders) | 1 (1) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Transamintis (Investigations) | 0 (0) | 8 (8)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Right thumb ischemia (Vascular disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 9 (9)
Epstein-Barr Virus (Infections and infestations) | 0 (0) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Creatinine Increase (Investigations) | 0 (0) | 5 (5)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased Phosphorous (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Swelling (General disorders) | 0 (0) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
edema (General disorders) | 0 (0) | 1 (1)
erythmea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT02385110/Prot_SAP_000.pdf